CLINICAL TRIAL: NCT05945602
Title: Optimization of Neurophysiologic Biomarkers for Rehabilitation Interventions in Veterans With Chronic Psychosis
Brief Title: Neurophysiologic Biomarkers for Cognitive Rehabilitation
Status: Recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: D4570-W; IK2RX004570 (NIH)
Record Dates: First submitted 2023-07-06; First posted 2023-07-14 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Schizophrenia Spectrum Disorders
Keywords: Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorde; Mental Disorders
MeSH Terms: conditions — Schizophrenia; Mental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Electrophysiological Recordings
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Biomarker Optimization - Patients: Veterans currently enrolled for healthcare services at the VA San Diego Healthcare System who have a diagnosis of a chronic psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
  Interventions: Other: Neurophysiologic Biomarker Assessments
- Biomarker Optimization - Healthy Comparison Subjects: Veterans currently enrolled for healthcare services at the VA San Diego Healthcare System who have no history of mental illness.
  Interventions: Other: Neurophysiologic Biomarker Assessments
- Biomarker Validation in Chronic Psychotic Disorders: Veterans currently enrolled for healthcare services at the VA San Diego Healthcare System with a diagnosis of a chronic psychotic disorder (e.g., schizophrenia or schizoaffective disorder).
  Interventions: Other: Neurophysiologic Biomarker Assessments

INTERVENTIONS:
Other: Neurophysiologic Biomarker Assessments — Non-invasive electroencephalography will be recorded to derive neurophysiologic biomarkers.

SUMMARY:
Cognitive symptoms of schizophrenia interfere with daily life-from managing self-care, to more complex tasks like taking medications and living independently. Unfortunately, these cognitive symptoms are not corrected by 'standard of care' treatments (antipsychotic medications), although some schizophrenia patients may experience modest clinical and cognitive benefits from cognitive remediation. To enhance the clinical impact of cognitive remediation and other rehabilitative interventions for Veterans living with chronic psychosis, this study will develop novel brain-based tools to help identify those Veterans who are most likely to benefit from pro-cognitive therapies. These studies may advance predictive algorithms that improve functional outcomes and life quality in Veterans with schizophrenia.

DETAILED DESCRIPTION:
This is an observational study recruiting Veterans with a diagnosis of Schizophrenia (SZ) and other Chronic Psychotic Disorders and Veterans in good general health (HS) who are enrolled in and/or receiving care at the VA San Diego Healthcare System. Eighty Veterans will undergo comprehensive neurophysiological, clinical, cognitive, and functional assessments in two "phases" (Phase 1: 30 SZ, 20 HS; Phase 2: 30 SZ).

In Phase 1 (Biomarker Optimization; Aims 1 & 2), Veterans will undergo systematic neurophysiologic testing designed to elicit spectral biomarkers linked to cortical excitation and inhibition ("E/I balance") during passive and stimulated conditions on two separate test visits (1-2 weeks apart). Experimental conditions will then be optimized for internal consistency and test-retest reliability using Generalizability Theory. The optimized biomarkers will be carried forward into Phase 2 (Biomarker Validation; Aim 3), where these neurophysiologic measures will be assessed before and after Veterans with SZ undergo 1 hour of cognitive training as a demonstration of neural system target engagement.

This proposal has 3 specific aims:

Aim 1. Identify the experimental conditions that optimize the psychometric properties (i.e., sensitivity to detect individual differences) of the spectral biomarkers linked to E/I balance.

Aim 2. Characterize the relationships of spectral biomarkers with rehabilitation-relevant outcomes.

Aim 3. Evaluate the sensitivity of the optimized E/I measures in predicting performance during an acute, 1-hour exposure to computerized cognitive training.

ELIGIBILITY:
Inclusion Criteria:

1. Have a DSM-5 diagnosis of a chronic psychotic disorder (e.g., schizophrenia, schizoaffective disorder, or delusional disorder); or b) are in good general mental and physical health (i.e., no active mental health condition).
2. Fluent in spoken and written English.
3. No impairment in hearing or vision.

Exclusion Criteria:

1. Active substance other than cannabis within the last 30 days as determined by self-report or positive urine toxicology (obtained as part of the screening process).
2. History of significant medical or neurological illness or intellectual disability.
3. Inability to comprehend or provide informed consent.
4. Specific to healthy comparison subjects: past or present diagnosis of schizophrenia, schizoaffective disorder, or other chronic psychotic disorder.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Veterans who are enrolled in and/or receiving healthcare services at the VA San Diego Healthcare System.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
1-week psychometric reliability of Aperiodic Spectral Biomarkers (neurophysiologic biomarker) | Approximately 7 days
  Estimates of aperiodic activity will be calculated from electroencephalography recordings collected at baseline (Day 1) and approximately 7 days later.

SECONDARY OUTCOMES:
Cognitive training performance | Day 1/ Baseline
  Performance on a computerized cognitive training exercise (i.e., the "Sound Sweeps" exercise) assessing auditory processing speed. Scores range between 0-1000, with greater scores indicating worse performance.
Cognition | Day 1/ Baseline
  Performance on MATRICS Consensus Cognitive Battery (MCCB). MCCB performance will be evaluated based on age- and gender-corrected T-scores (normative mean = 50; standard deviation = 10). Higher T-score values indicate better performance.
Symptoms | 1 visit
  Scores on the Positive and Negative Syndrome Scale (PANSS)
Functioning | Day 1/ Baseline
  Scores on the World Health Organization Disability Assessment Schedule (WHODAS 2.0). WHODAS summary scores are converted into a metric ranging from 0 to 100 (where 0 = no disability; 100 = full disability).
Functioning - Quality of Life | Day 1/ Baseline
  Scores on the World Health Organization Quality of Life Scale (WHOQOL-BREF). WHOQOL-BREF domain scores are converted into a metric ranging from 0 to 100 (where 0 = very poor quality of life; 100 = very good quality of life).

CONTACTS AND LOCATIONS:
Overall Officials: Juan Molina, MD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No